CLINICAL TRIAL: NCT03591679
Title: Role of Bilateral Uterine Artery Ligation in Reducing Incidence of Postpartum Hemorrhage in Cesarean Section in Patients At Risk of Uterine Atony A Randomized Controlled Trial
Brief Title: Bilateral Uterine Artery Ligation in Reducing Incidence of Postpartum Hemorrhage in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUALCS
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients at risk of uterine atony undergoing cesarean section underwent bilateral uterine artery ligation and received oxytocin.
  Interventions: Drug: Oxytocin; Procedure: bilateral uterine artery ligation
- control group (Active Comparator): patients at risk of uterine atony undergoing cesarean section received oxytocin only.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 20 units by slow intravenous drip injection
Procedure: bilateral uterine artery ligation — • The peritoneum over the vesico-uterine pouch already being incised horizontally, the peritoneum over the uterine isthmus and cervix was dissected downwards, and this dissection was then extended laterally.
  Arms: study group

SUMMARY:
The patients were recruited from women attending labor ward to undergo cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women with one or more of the following conditions undergoing cesarean section for obstetric indication were included:
* Maternal anemia (not less than 7 gm %).
* Macrosomic baby >4kgs.
* Twin pregnancy and high order pregnancy.
* Polyhydramnios.
* Grand multipara.
* Previous history of atonic postpartum hemorrhage.
* Prolonged vaginal delivery.
* Emergency cesarean.
* Chorioamnionitis.

Exclusion Criteria:

* - Placenta previa.
* Patients with bleeding tendency (congenital or acquired)
* Ante-partum hemorrhage.
* Patients with no risk for uterine atony.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
mean Blood loss after placental separation | 30 minutes
  by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Samy A, Ali MK, Abbas AM, Wahab HA, Wali AA, Hussien AH, Mostafa M, Taymour MA, Ogila AI, Ahmad Y, Essam A, Mahmoud M. Randomized controlled trial of the effect of bilateral uterine artery ligation during cesarean among women at risk of uterine atony. Int J Gynaecol Obstet. 2020 Feb;148(2):219-224. doi: 10.1002/ijgo.13064. Epub 2019 Dec 10. PMID 31755559